CLINICAL TRIAL: NCT00000953
Title: Evaluation of Brovavir ( BV-ara-U; SQ 32,756 ) Versus Acyclovir in the Treatment of Localized Herpes Zoster in HIV-Infected Patients
Brief Title: Comparison of Brovavir Versus Acyclovir in the Treatment of Herpes in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); Glaxo Wellcome (Industry)
Purpose: Treatment
Other Study IDs: ACTG 169; Protocol -38/-022
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections; Chickenpox
Keywords: Herpes Zoster; Acyclovir; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; sorivudine
MeSH Terms: conditions — HIV Infections; Chickenpox; Herpes Zoster; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — sorivudine; Acyclovir

INTERVENTIONS:
Drug: Sorivudine
Drug: Acyclovir

SUMMARY:
To compare the efficacy of oral sorivudine (brovavir) and oral acyclovir for the treatment of localized herpes zoster in HIV-infected patients.

HIV-infected patients are at high risk for herpesvirus infections, including varicella-zoster virus ( VZV ) infections, also called shingles. Acyclovir, an approved drug, is widely used to treat VZV infections in the HIV population. Since no data from controlled studies are available to define the role of antiviral therapy for VZV infections in HIV-infected patients, a study is needed to test the relative efficacy of brovavir, an experimental antiviral drug, versus that of acyclovir.

DETAILED DESCRIPTION:
HIV-infected patients are at high risk for herpesvirus infections, including varicella-zoster virus ( VZV ) infections, also called shingles. Acyclovir, an approved drug, is widely used to treat VZV infections in the HIV population. Since no data from controlled studies are available to define the role of antiviral therapy for VZV infections in HIV-infected patients, a study is needed to test the relative efficacy of brovavir, an experimental antiviral drug, versus that of acyclovir.

One hundred-eighty patients are randomized to receive either brovavir or acyclovir as follows: brovavir or its matching placebo once daily and acyclovir or its matching placebo five times daily. Treatment continues for 10 days. Entry into the study must occur within 72 hours of lesion development. Patients are followed in person daily or at regular intervals during study drug administration and on days 14, 21, and 28, and then monthly by telephone for 11 months thereafter.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Medication for concurrent conditions (e.g., insulin, antihypertensives, bronchodilators, digoxin) or antibacterials or antifungals to treat concurrent infections at other sites or superinfection of the zoster lesion.
* Anti-inflammatory, analgesic (including narcotic analgesic), or antipyretic agents.
* Antidepressants and antipsychotics such as amitriptyline and/or fluphenazine.
* Nerve blocks.
* AZT, ddI, ddC, and amantadine.
* Low-dose corticosteroids for treatment of an underlying (not zoster-related) disease.
* Immune modulators without varicella-zoster virus activity (e.g., GM-CSF, gp160 vaccine).

Patients must have:

* HIV infection.
* Localized, cutaneous herpes zoster (shingles).
* Zoster-associated rash present for 3 or fewer days prior to entry.

Prior Medication:

Allowed:

* Zidovudine.
* ddI.
* ddC.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions and symptoms are excluded:

* Chickenpox.
* Evidence of visceral dissemination (organ involvement, i.e., brain, liver, or lung) and/or cutaneous dissemination (more than 20 vesicles in dermatomes beyond contiguous dermatomes) of zoster.
* Zoster-like lesion caused by organism other than VZV (e.g., HSV, enterovirus, or Mycoplasma).
* Bacterial superinfection of zoster lesion.
* Zosteriform lesion previously treated with topical antiviral agents.
* Acute, life-threatening opportunistic infection requiring treatment (ongoing suppressive or prophylactic maintenance therapy other than ganciclovir or foscarnet is permitted).
* Concurrent severe disease that may either impair ability to take oral medication in capsule or tablet form or limit survival during the 10-day treatment period or during acute phase follow-up (28 days).
* Suspected acute deterioration of renal or hepatic function.
* Mental impairment that precludes ability to comply with protocol.
* Any condition that would render the patient unsuitable for treatment.

Concurrent Medication:

Excluded during acute phase of study:

* Antiviral medications other than AZT, ddI, ddC, or anti-Parkinson's drugs (i.e., amantadine).
* Interferon.
* Isoprinosine.
* Levamisole.
* Transfer factor.
* Topical virucidal agents, oxidizing agents, DMSO, cell division-stimulating/healing agents, or astringents.
* Topical anesthetics (such as capsaicin or xylocaine).
* Topical creams or ointments that may interfere with evaluation of zoster lesions.
* Cimetidine.
* Fluorouracil or its derivatives, flucytosine, or cyclophosphamide (during drug administration and for 2 weeks thereafter).
* High-dose corticosteroids.
* Anticoagulant therapy (heparin locks and low-dose warfarin sodium permitted).
* Probenecid or derivatives.
* Treatment for any acute, life-threatening opportunistic infection (suppressive or prophylactic maintenance therapy other than ganciclovir or foscarnet is permitted).

Use of the following drugs is discouraged during the long-term phase of the study:

* Antiviral agents with VZV activity.
* Immunomodulators with presumed VZV activity.
* VZV immune globulin.
* Capsaicin.
* Cimetidine.

Patients with the following prior conditions are excluded:

* History of immediate hypersensitivity or serum sickness reaction or idiosyncratic reaction (such as hepatic necrosis or Stevens-Johnson syndrome) to any nucleoside analog antiviral agent or to any anticancer therapy with cytolytic agents.

Prior Medication:

Excluded within 1 month prior to entry:

* Any investigational drugs or treatments not licensed for any indication (other than ddI or ddC).

Excluded within 2 weeks prior to entry:

* Any systemic antiviral therapy, including ganciclovir, foscarnet, vidarabine, acyclovir, or ribavirin.
* Any antiretroviral drug other than zidovudine, ddI, and ddC.
* Immune globulin (e.g., IgG, VZIG).

Excluded within 72 hours prior to entry:

* Cyclophosphamide.
* Flucytosine.
* Fluorouracil or its derivatives.

Alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Primary Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crumpacker C, Study Chair
Locations (44):
- United States (44):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA Med Ctr, Los Angeles, California
  - Veterans Administration Med Ctr, Martinez, California
  - Infectious Disease Med Group, Oakland, California
  - San Diego Naval Hosp, San Diego, California
  - Mount Zion Med Ctr, San Francisco, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Veterans Administration Med Ctr / Community AIDS Program, Washington D.C., District of Columbia
  - Med College of Georgia, Augusta, Georgia
  - Univ of Hawaii / Leahi Hosp, Honolulu, Hawaii
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Natl Institutes of Health / NIAID, Bethesda, Maryland
  - Massachusetts Gen Hosp / Harvard Med School, Boston, Massachusetts
  - Beth Israel Hosp, Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - New England Deaconess Hosp, Boston, Massachusetts
  - Washington Univ, St Louis, Missouri
  - Univ of New Mexico, Albuquerque, New Mexico
  - Beth Israel Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - SUNY / Health Sciences Ctr at Stony Brook, Stony Brook, New York
  - SUNY / Health Sciences Ctr at Syracuse, Syracuse, New York
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Univ Dermatology Associates, Cincinnati, Ohio
  - Ohio State Univ / ACTU-Univ Clinic, Columbus, Ohio
  - Dayton Veterans Administration Med Ctr, Dayton, Ohio
  - Med College of Ohio, Toledo, Ohio
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Dallas Veterans Administration Med Ctr, Dallas, Texas
  - Univ of Texas, Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Univ TX San Antonio Health Science Ctr, San Antonio, Texas
  - Scott and White Hosp, Temple, Texas
  - Univ of Virginia Health Sciences Ctr, Charlottesville, Virginia
  - Virginia Clinical Research Inc, Norfolk, Virginia
  - Salem Veterans Administration Med Ctr, Salem, Virginia
  - Univ of Washington, Seattle, Washington
  - Great Lakes Hemophilia Foundation, Wauwatosa, Wisconsin

REFERENCES:
- [Background] Gnann J, et al. Sorivudine (BV-araU) versus acyclovir for Herpes zoster in HIV-infected patients. Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:55